CLINICAL TRIAL: NCT03916770
Title: The Effect of Whole Body Vibration on Spasticity in Poststroke Hemiplegia:Prospective Randomized Controlled Research
Brief Title: The Effect of Whole Body Vibration (WBV) on Spasticity in Poststroke Hemiplegia
Acronym: WBV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstPMRTRH-BMR
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Muscle Spasticity; Physiology
Keywords: muscle; vibration; H reflex; H/M ratio; spasticity
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: Whole Body Vibration (WBV) will be applied to Poststroke Hemiplegia. The patients are divided in two groups; WBV group and shame WBV group.
Who Masked: Participant
Masking Description: Patients will be blind to treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- whole body vibration (Active Comparator): WBV(whole body vibration) will be applied to interventional group for 4 weeks, 3 days a week, a total of 12 sessions while standing upright with the WBV powerplate pro5 device.(Vibration frequency: 30Hz, amplitude: 2.2 mm at progressively increasing duration)
  Interventions: Device: Real vibrator
- Sham whole body vibration (Sham Comparator): The sham WBV will be applied to the Control group. A WBV device with 99.5% weakened amplitude will be used for sham WBV. (Application duration of the sham WBV will be same as WBV in the treatment group ).
  Interventions: Device: Sham vibrator

INTERVENTIONS:
Device: Sham vibrator — The Sham control group will have WBV the same time,in the same position with the same frequency but 99.5% weakened amplitude.
  Other Names: Sham WBV
  Arms: Sham whole body vibration
Device: Real vibrator — The intervention group will have WBV(frequency:30Hz,amplitude:2,2mm,at upright position
  Other Names: Real WBV
  Arms: whole body vibration

SUMMARY:
The primary purpose of this study is to show whether WBV application has antispastic effect. The secondary aim is to demonstrate whether WBV has neuromodulatory activity on increased stretch reflex and motor neuron activity, which is the basis of the pathophysiology of spasticity.Hypotheses of this study:Whole body vibration in poststroke hemiplegia reduces ankle plantar flexion spasticity.

1. WBV ; reduces plantar flexor spasticity after stroke
2. WBV decreases poststroke spasticity, by decreasing increased stretch reflex and motor neuron activity.

DETAILED DESCRIPTION:
Patients with a stroke of at least 1 month before and with a history of ankle plantar flexion spasticity will be included in the study. Conventional rehabilitation program will be applied to all patients (n=48).The intervention group (n=24) will be applied for 4 weeks, 3days a week, a total of 12 sessions with the WBV powerplate pro5 device. In the WBV group, the frequency and acceleration of vibration will be 30Hz and 18.0m/s2, respectively. The WBV exercise intensity will progressively increase throughout the twelve-session. In the control group, the same procedures will be followed. However, unlike the WBV group, a vibration will be given whose acceleration is attenuated by 99.5%.The surface Electromyography (EMG) and degree of spasticity of soleus muscle will be evaluated at the beginning and end of the all sessions. Soleus H-reflex will be recorded with surface EMG.To obtain the H-reflex response, the posterior tibial nerve in the popliteal region will be stimulated by using a stimulator (FE155 Stimulator HC ADInstrument, Oxford UK) with 1 ms-pulse current. The records will be taken with the Ag / AgCl electrodes (Kendall ®Coviden, self-adhesive electrodes) placed on skin according to the SENIAM protocol. The degree of spasticity will be measured as a soleus muscle tone torque on a fixed angular velocity moving platform.The data will be recorded with the PowerLab data acquisition device

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic / hemorrhagic poststroke hemiplegia aged 18-90 years,
2. Stroke time ≥1 months,
3. Ankle plantar flexor spasticity MAS ≥1,
4. Brunnstrom stage ≥3 for lower extremity,
5. Patients who were standing for more than five minutes and had a static balance

Exclusion Criteria:

1. Cardiac disorder (rhythm / conduction disorder, cardiac pacemaker, ischemic heart disease)
2. Lower extremity fracture,
3. Findings or suspicion of active deep vein thrombosis,
4. A history of deep vein thrombosis and pulmonary embolism,
5. Orthostatic hypotension
6. Resistant hypertension,
7. Peripheral nerve lesions such as polyneuropathy, radiculopathy
8. Active inflammatory, rheumatologic or infectious disease,
9. Ankle,knee or hip joint contracture,
10. Presence of panic attacks,
11. Patients with dizziness and balance problems,
12. Patients with not intact skin surface to connect electrodes
13. Patients with communication problems: aphasia, major depression
14. Epilepsy
15. Patients who received botulinum A toxin in the last 6 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
spasticity-torque | 4 weeks
  Spasticity will be measured as a torque. The unit is Nm
spasiticity-modified Ashworth scale | 4 weeks
  The spasticity degree of the plantar flexors will be evaluated by using a subjective assessment method (modified Ashworth scale-MAS)
spasticity-homosynaptic post-activation depression (HPAD) | 4 weeks
  Homosynaptic post-activation depression is a presynaptic mechanism regulating the excitability of the stretch reflex. Decreased presynaptic inhibition and homosynaptic depression are also thought to play a role in the pathophysiology of spasticity. The higher HPAD, the lower spasticity
Motor neuron activity-Hmax / Mmax ratio | 4 weeks
  Hmax / Mmax ratio defines motor neuron activity. The higher this ratio, the higher the activity of motor neuron pool

CONTACTS AND LOCATIONS:
Overall Officials: Ayşenur Bardak, Prof, Study Chair — Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital Istanbul, Turkey, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan KS, Liu CW, Chen TW, Weng MC, Huang MH, Chen CH. Effects of a single session of whole body vibration on ankle plantarflexion spasticity and gait performance in patients with chronic stroke: a randomized controlled trial. Clin Rehabil. 2012 Dec;26(12):1087-95. doi: 10.1177/0269215512446314. Epub 2012 Oct 3. PMID 23035004
- [Background] Pang MY, Lau RW, Yip SP. The effects of whole-body vibration therapy on bone turnover, muscle strength, motor function, and spasticity in chronic stroke: a randomized controlled trial. Eur J Phys Rehabil Med. 2013 Aug;49(4):439-50. Epub 2013 Mar 13. PMID 23486302
- [Background] Miyara K, Matsumoto S, Uema T, Noma T, Ikeda K, Ohwatashi A, Kiyama R, Shimodozono M. Effect of whole body vibration on spasticity in hemiplegic legs of patients with stroke. Top Stroke Rehabil. 2018 Mar;25(2):90-95. doi: 10.1080/10749357.2017.1389055. Epub 2017 Oct 16. PMID 29032720
- [Background] Brogardh C, Flansbjer UB, Lexell J. No specific effect of whole-body vibration training in chronic stroke: a double-blind randomized controlled study. Arch Phys Med Rehabil. 2012 Feb;93(2):253-8. doi: 10.1016/j.apmr.2011.09.005. PMID 22289234
- [Background] Alp A, Efe B, Adali M, Bilgic A, Demir Ture S, Coskun S, Karabulut M, Ertem U, Gunay SM. The Impact of Whole Body Vibration Therapy on Spasticity and Disability of the Patients with Poststroke Hemiplegia. Rehabil Res Pract. 2018 May 2;2018:8637573. doi: 10.1155/2018/8637573. eCollection 2018. PMID 30225145